CLINICAL TRIAL: NCT00117351
Title: A Multicenter, Open-Label, Phase 2 Study of VELCADE (Bortezomib) for Injection in Previously Treated Patients With Stage IIIB and IV Bronchioloalveolar Carcinoma and Adenocarcinoma With Bronchioloalveolar Features
Brief Title: VELCADE in Previously Treated Patients With Stage IIIB and IV Bronchioloalveolar Carcinoma (BAC) and Adenocarcinoma With BAC Features
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient efficacy
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05002; NCT00119223 (obsolete NCT alias)
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar
Keywords: Adenocarcinoma; Bronchiolo-Alveolar; Carcinoma, Bronchioloalveolar; Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchiolo-Alveolar
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma | interventions — Bortezomib

INTERVENTIONS:
Drug: VELCADE

SUMMARY:
This study will evaluate the safety and efficacy of VELCADE in patients with previously treated stage IIIB and IV bronchioloalveolar carcinoma and adenocarcinoma with bronchioloalveolar features.

DETAILED DESCRIPTION:
Bronchioloalveolar carcinoma (BAC) and adenocarcinoma with bronchioloalveolar features are distinct subtypes of non-small-cell lung cancer which are difficult to treat in advanced stages. This study will determine the safety and efficacy of VELCADE therapy in patients with advanced BAC or adenocarcinoma with BAC features who have failed epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed BAC or adenocarcinoma with BAC features.
* Have stage IIIB (malignant pleural effusion) or stage IV disease.
* Have progressed on or after receipt of 1 to 2 prior lines of chemotherapy, one of which must be an EGFR TKI (Iressa or Tarceva). Adjuvant chemotherapy will NOT be counted as a prior line of therapy.
* Have radiographic documentation of progressive disease (PD) as determined by the investigator.
* Have measurable disease by RECIST.
* Are 18 years of age or older.
* Have a life expectancy greater than 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Are able to provide written informed consent in accordance with all applicable regulations and follow the study procedures.
* Patients must be capable of understanding the investigational nature and potential risks and benefits.

Exclusion Criteria:

* Have had chemotherapy (or an EGFR TKI) 4 weeks prior to enrollment.
* Have peripheral neuropathy of Grade 2 or greater intensity, as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 3.0).
* Have been previously treated with VELCADE.
* Have experienced myocardial infarction within 6 months prior to enrollment or have New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Have had radiation therapy within 4 weeks prior to enrollment.
* Have had monoclonal antibody therapy within 4 weeks prior to enrollment.
* Have had any major surgery within 4 weeks prior to enrollment.
* Have inadequate organ function at the Screening visit as defined by laboratory testing
* Have symptomatic brain metastases or brain metastases that have not responded to radiation therapy, local or systemic chemotherapy, or were not completely resected by stereotactic surgery or other surgical modalities, or have significant post treatment brain edema.
* Have uncontrolled active systemic infection requiring treatment.
* Have had treatment for a cancer other than BAC within 5 years prior to enrollment, with the exception of basal cell carcinoma or cervical cancer in situ.
* Have a history of allergic reaction attributable to compounds containing boron or mannitol or hypersensitivity reactions to drugs formulated with polysorbate 80.
* Have known human immunodeficiency virus (HIV)-positive or hepatitis B surface antigen-positive status or known active hepatitis C infection. Patients assessed by the investigator to be at risk for HIV, hepatitis B or C infection should be tested in accordance with local regulations.
* Have poorly controlled hypertension, diabetes mellitus, or another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Are a pregnant or breast-feeding female. Confirmation that the patient is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during the screening period. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Are unwilling to employ adequate means of contraception (condoms, diaphragm, birth control pills, injections, intrauterine device, or abstinence).
* Are currently receiving or have previously received an investigational agent for any reason within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States